CLINICAL TRIAL: NCT00761033
Title: Music to Reduce Pain and Anxiety in the Pediatric Emergency Department: a Randomized Controlled Trial of Children 3-6 Years Undergoing Intravenous Placement
Brief Title: Music to Reduce Pain and Anxiety in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Stollery Children's Hospital Foundation (Other)
Responsible Party: Lisa Hartling/Assistant Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-010908
Record Dates: First submitted 2008-09-25; First posted 2008-09-26 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Pain; Distress
Keywords: children undergoing intravenous placement in the pediatric emergency department
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- music (Experimental): children will listen to music during procedure
  Interventions: Behavioral: music
- Standard care (Other): Standard care
  Interventions: Behavioral: music

INTERVENTIONS:
Behavioral: music

SUMMARY:
Many medical procedures aimed at helping children can cause them pain and distress. If children experience certain levels of pain or distress, it can have long lasting negative effects. The emergency department can be a particularly stressful place for children and their parents. There are also many procedures that children may have in the emergency department that can cause pain and distress. These include procedures such as needle pokes, stitches, or setting a broken bone. Two common methods of managing a child's pain in the emergency department are drugs and distraction. Drugs are not always practical and may come with unwanted side effects. Distraction is often used formally or informally and by parents or the health professionals. One form of distraction involves listening to music. This can lower the child's pain and distress by moving their attention from the painful stimulus, for example a needle poke, to a more pleasant sensation such as familiar children's songs. This study will test whether music is useful to help lower pain and distress for young children (ages 3 to 6 years) who are visiting an emergency department and need an intravenous line. Music is safe and pleasant for children. The results from this study could be important for many children receiving medical care.

ELIGIBILITY:
Inclusion Criteria:

* Children attending the pediatric ED between the ages of 3 and 6 years - Undergoing an IV placement
* Conscious
* Have sufficient knowledge of the English language to understand and follow instructions and complete the age-appropriate pain assessment

Exclusion Criteria:

* Children with hearing impairments, developmental disabilities, or sensory impairment to pain (e.g., spina bifida)
* Children will be excluded at the discretion of the attending staff (e.g., child in critical condition; requires urgent IV placement; or has altered level of consciousness).

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Estimated)
Dates: Start 2008-10

PRIMARY OUTCOMES:
Observation Scale of Behavioral Distress-Revised (OSBD-R)

SECONDARY OUTCOMES:
Pain

CONTACTS AND LOCATIONS:
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

REFERENCES:
- [Result] Hartling L, Newton AS, Liang Y, Jou H, Hewson K, Klassen TP, Curtis S. Music to reduce pain and distress in the pediatric emergency department: a randomized clinical trial. JAMA Pediatr. 2013 Sep;167(9):826-35. doi: 10.1001/jamapediatrics.2013.200. PMID 23857075